CLINICAL TRIAL: NCT05189743
Title: A Prospective Multi-centre Randomised Study for Treatment of Burns With Dermis Graft or Split-thickness Skin Auto-graft.
Brief Title: The Dermisgraft Epithelialization and Late Scar Healing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Folke Sjoberg, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2.4
Record Dates: First submitted 2021-11-18; First posted 2022-01-12 (Actual); Last update posted 2022-01-12 (Actual); Status verified 2021-12

CONDITIONS: Burns
MeSH Terms: conditions — Burns

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dermis graft (Experimental)
  Interventions: Procedure: Skin transplantation to heal burn injuries
- STSG (Experimental)
  Interventions: Procedure: Skin transplantation to heal burn injuries

INTERVENTIONS:
Procedure: Skin transplantation to heal burn injuries — The study compare two different treatment modalities, STSG (split-thickness skin graft) versus dermis graft after excision of devitalized/necrotic tissue.
  A dermatome will be used for graft harvest.

SUMMARY:
Study Synopsis

Title; The dermis graft: epithelialization and late scar evaluation A Clinical Prospective multicenter trial

Objectives; The objective of this study is to compare a dermal graft with a conventional split thickness skin graft regarding healing quality and scarring.

Design; the study is a prospective, controlled clinical multicenter trial.

Study population; Atleast 20 burn patients (18-80 years) with a full thickness burn that requires permanent skin cover.

Time plan; Enrollment will continue until atleast 20 patients have been included and completed the study.

DETAILED DESCRIPTION:
Background: Donor site morbidity is a major concern such as wound healing disturbances, hypertrophic scarring and hypo-/hyperpigmentation. The dermal graft technique is an alternative to the standard split-thickness skin graft (STSG) technique to minimize donor site morbidity. Immediate cover of the donor site after harvest leaving a non-exposed wound is a big advantage. The aim of the study was to compare the functional and aesthetic outcome between two treatment methods (dermal graft with STSG).

Methods: From February 2017 to December 2020, 21 patients received a dermis graft and a regular split-thickness skin graft in a prospective randomized study design. The recipient and the donor site were compared separately regarding healing time, scarring and patient subjective satisfaction. All sites (both donor and recipient) were analyzed histologically regarding remodeling and scar formation.

ELIGIBILITY:
Inclusion Criteria:

* Thermal & chemical burns < 30 % TBSA
* Males & females between 18-80 years old
* At least one coherent full thickness wound measuring 15 x 7.5 cm
* A minimal of 15 x 7.5 cm coherent undamaged skin located at frontal or lateral side of one of the thighs for graft harvest.

Exclusion Criteria:

* Patients with severe cutaneous trauma at the same site as the burn injury
* Previous burns at the treatment site
* Severe cognitive dysfunction or psychiatric disorder
* Chronic skin disorder
* Chronic use of systemic or local corticosteroid
* Chronic use of anticoagulants or platelets
* Autoimmune disease
* Active hepatitis
* Full thickness burns of head, genitalia, axilla or upper third of medial upper arm

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Healing time | 4 weeks
  Recipient sites are to be assessed regarding healing (re-epithelization) at each site (donor respective recipient). Healing will be assesed in days after surgery.
Aesthetic outcome | 12 months
  The aesthetic appereance regarding scarring will be assessed. A MPA580 cutometer will asses the viscoelasticity in the skin and POSAS will asses the appereance of the scar objectively as subjectively.
  R0 and R2 will be used as variables evaluating firmness and elasticity.
  POSAS will be analysed accoring to a scoring system (0-10 and 0-60).

CONTACTS AND LOCATIONS:
Locations (1):
- Linköpings Unversity Hospital, Linköping, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Derived] Dogan S, Elmasry M, El-Serafi A, Sjoberg F, Vuola J, Kankuri E, Grigoriadi MP, Valtonen J, Abdelrahman I, Steinvall I, Karlsson M, Olofsson P, Lindford A. A prospective dual-centre intra-individual controlled study for the treatment of burns comparing dermis graft with split-thickness skin auto-graft. Sci Rep. 2022 Dec 15;12(1):21666. doi: 10.1038/s41598-022-25346-4. PMID 36522434